CLINICAL TRIAL: NCT00122629
Title: Triple Therapy With Peg-Interferon Alfa-2b/Ribavirin Plus Amantadine Compared to Standard Peg-Interferon Alfa-2b/Ribavirin for Previous HCV Non Responders ANRSHC03 BITRI
Brief Title: Triple Therapy With Peg-Interferon Alfa-2b/Ribavirin Plus Amantadine Compared to Standard Peg-Interferon Alfa-2b/Ribavirin for Previous Hepatitis C Virus (HCV) Non Responders
Status: Terminated | Phase: Phase 3 | Type: Interventional
Sponsor: French National Agency for Research on AIDS and Viral Hepatitis (Other Government)
Collaborators: Schering-Plough (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ANRSHC03 BITRI
Record Dates: First submitted 2005-07-20; First posted 2005-07-22 (Estimated); Last update posted 2005-07-29 (Estimated); Status verified 2005-07

CONDITIONS: Hepatitis C, Chronic
Keywords: Hepatitis C, Chronic; peginterferon alfa-2b; ribavirin; Amantadine
MeSH Terms: conditions — Hepatitis C, Chronic | interventions — peginterferon alfa-2b; Ribavirin; Amantadine

INTERVENTIONS:
Drug: peg-interferon alfa-2b
Drug: ribavirin
Drug: amantadine

SUMMARY:
Triple antiviral therapy with peg-interferon-alfa/ribavirin+amantadine was suggested to increase sustained virological response (SVR) rates in HCV non-responders to a standard interferon/ribavirin combination.

Patients with hepatitis C virus infection were eligible if they had failed to respond to a single previous 24 week cycle of interferon/ribavirin combination therapy. Non-response was defined as persistent HCV RNA in the serum during the last month of treatment.

This study tested the efficacy and safety of pegylated interferon alfa-2b with ribavirin and amantadine or a placebo for 48 weeks.

DETAILED DESCRIPTION:
Triple antiviral therapy with peg-interferon-alfa/ribavirin + amantadine was suggested to increase sustained virological response (SVR) rates in HCV non-responders to a standard interferon/ribavirin combination.

The aim of this study is to determine if the addition of amantadine to PEG-IFN/ribavirin enhances SVR.

This study is a double blind, comparative, prospective multicenter, randomized study. Patients are recruited from 23 hepatology centers in France. The protocol was approved by the French ethical committee and all patients provided written informed consent. Eligible subjects are randomly assigned to the two treatment groups in equal proportions. The randomization process is generated by the Department of Biostatistics, Hospices Civils de Lyon, Lyon, France.

Main inclusion criteria are: elevated ALT, detectable HCV RNA, Metavir score over or equal to A1F1 and below or equal to F3. Patients received PEG-IFN 1.5µg/kg/week, ribavirin 800-1200mg/day and amantadine 200mg/day or placebo during 48 weeks.

The primary endpoint is a sustained virological response, defined as an undetectable HCV-RNA 24 weeks after treatment discontinuation (week 72). Secondary endpoints are the biochemical response at week 72 defined as ALT normalization; histological benefit; tolerance; and virological and biochemical responses during therapy at weeks 12, 24 and 48.

ELIGIBILITY:
Inclusion Criteria:

* Positive anti-HCV antibody test
* Patients who did not respond to treatment with standard interferon + ribavirin (HCV RNA+ by PCR in the last month of treatment)
* Compensated liver disease
* Neutrophil count over or equal to1000/mm3
* Platelet count over or equal to 100 giga/L
* Haemoglobin over or equal to 10g/dL
* Patients had to have undergone a post-treatment liver biopsy within a year, showing a METAVIR histological score over or equal to A1F1, without cirrhosis (fibrosis score below F4)
* ALT over N and HCV RNA+ at screening

Exclusion Criteria:

* Co-infection with hepatitis B or human immunodeficiency virus
* Any other cause of liver disease
* Active drug abuse, active alcohol consumption above 40g/day
* Organ grafts
* Presence of hepatocellular carcinoma
* Cardiovascular, metabolic, renal, haematological, neurological or psychiatric disease
* Patients with previous amantadine use
* Systemic immunosuppressive or antiviral treatment during the last 24 weeks and those with a history of interferon and/or ribavirin intolerance

Ages: 18 Years to 65 Years | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 405
Dates: Start 2000-10; Study Completion 2003-05

PRIMARY OUTCOMES:
Sustained virological response, defined as an undetectable HCV-RNA 24 weeks after treatment discontinuation at week 72

SECONDARY OUTCOMES:
Biochemical response at week 72 defined as ALT normalization
Histological benefit
Tolerance
Virological and biochemical responses during therapy at weeks 12, 24 and 48

CONTACTS AND LOCATIONS:
Overall Officials: Christian Trepo, MD, Principal Investigator — Hépato-Gastroentérologie Hopital Hôtel-Dieu LYON; P. ADELEINE, MD, Study Chair — Laboratoire d'Informatique Médicale Lyon
Locations (1):
- Service d'Hépato-Gastroentérologie Hopital Hotel Dieu, Lyon, France